CLINICAL TRIAL: NCT06925061
Title: A Phase 2 Multicentre, Randomised, Parallel-arm, Placebo-controlled, Double-blind Study to Evaluate the Safety and Target Engagement of EXL01 in the Prevention of Post-operative Recurrence of Crohn's Disease
Brief Title: Target Engagement of EXL01 in the Prevention of Post-operative Recurrence of Crohn's Disease
Acronym: MAINTAIN-POP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Madeleine Bezault (Other)
Responsible Party: Sponsor-Investigator, Madeleine Bezault, Principal investigator, Saint-Louis Hospital, Paris, France
Organization: Saint-Louis Hospital, Paris, France (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: REMIND_2024-001_EXL01; 2024-511357-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-30; First posted 2025-04-13 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease (CD)
MeSH Terms: conditions — Crohn Disease | interventions — Postoperative Period

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live biotherapeutic product (EXL01) (Experimental): EXL01 administered with or without SoC treatment orally, once a day during 24 weeks
  Interventions: Drug: After surgery for Crohn's disease, eligible patients will be randomized 1:1 to receive oral EXL01 or placebo with or without SoC treatment (based on investigator decision) for up to 24 weeks
- Placebo (Placebo Comparator): Placebo administered with or without SoC treatment orally, once a day during 24 weeks
  Interventions: Drug: After surgery for Crohn's disease, eligible patients will be randomized 1:1 to receive oral EXL01 or placebo with or without SoC treatment (based on investigator decision) for up to 24 weeks

INTERVENTIONS:
Drug: After surgery for Crohn's disease, eligible patients will be randomized 1:1 to receive oral EXL01 or placebo with or without SoC treatment (based on investigator decision) for up to 24 weeks — Randomisation will be stratified on post-surgical treatment (none vs anti-TNF), and on smoking status (non-smoker vs smoker).

SUMMARY:
MAINTAIN-POP is a Phase 2, randomised, double-blind, placebo-controlled, multicenter study of the impact of oral administration of EXL01 in the prevention of post-operative endoscopic recurrence of Crohn's disease after surgery.

Approximately 80 eligible patients will be randomized 1:1 to receive oral EXL01 or placebo with or without SoC treatment (based on investigator decision) for up to 24 weeks or until a study or treatment discontinuation criterion is met. Randomisation will be stratified on post-surgical treatment (none vs anti-TNF), and on smoking status (non-smoker vs smoker).

The primary objective is to compare the distribution of endoscopic modified Rutgeerts scores, as centrally assessed, at 6 months post-surgery in patients with CD treated with EXL01 to patients treated with placebo. Endoscopic recurrence will be assessed using the endoscopic score assessed by central reading at Week 24 after surgery. All participants will be followed for safety until 4 weeks after end of treatment.

DETAILED DESCRIPTION:
MAINTAIN-POP is a Phase 2, randomised, double-blind, placebo-controlled, multicenter study of the impact of oral administration of EXL01 in the prevention of post-operative endoscopic recurrence of Crohn's disease after surgery.

After surgery for Crohn's disease, as per institutional Standard of Care (SoC), approximately 80 eligible patients will be randomized 1:1 to receive oral EXL01 or placebo with or without SoC treatment (based on investigator decision) for up to 24 weeks or until a study or treatment discontinuation criterion is met. Randomisation will be stratified on post-surgical treatment (none vs anti-TNF), and on smoking status (non-smoker vs smoker).

The primary objective is to compare the distribution of endoscopic modified Rutgeerts scores, as centrally assessed, at 6 months post-surgery in patients with CD treated with EXL01 to patients treated with placebo.. All patients will be monitored continuously for safety while on the study treatment. Endoscopic recurrence will be assessed using the endoscopic score assessed by central reading at Week 24 after surgery. Faecal and blood samples for biomarker assessments will be obtained at Weeks 0, 4, 12, and 24. Patients who experience disease flare before Week 24 will discontinue the study treatment (EXL01 or placebo) and undergo an early discontinuation (ED) visit. All participants will be followed for safety until 4 weeks after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female aged ≥18 years at the time of providing documented informed consent.
* Has a diagnosis of CD with ileal involvement (ileal only or ileocolonic; L1 or L3 in Montreal classification) for at least 3 months prior to Screening.
* Has undergone an ileocecal resection or iterative ileo-colonic resection, as per institutional SoC, between 5 days to 5 weeks before randomization.
* Is scheduled, in SoC context, to receive no treatment for CD or anti-TNF agents in the 6 months after surgery

Exclusion Criteria:

* Has a not recovered adequately from any toxicity and/or complications from the surgery before the first dose of study intervention
* Has a current stoma. Inclusion will be possible after continuity restoration (during the 5 weeks following continuity restoration)
* Has active anal fistula
* Is scheduled, according to SoC, to receive a biotherapy at the exception of anti-TNF agent in the 6 months after surgery
* Has had more than 2 past small bowel resections or cumulated intestinal resection superior to 50 cm
* Has a contraindication to endoscopy or anaesthesia.
* Is receiving antibiotics at time of randomization or is likely to require antibiotic treatment within 6 weeks of the first dose of EXL01 or placebo.
* Has a history of hypersensitivity to EXL01 and/or any excipients, which are listed in the Investigator Brochure (IB), and/or to soybean or soy-containing products.
* Has a not recovered adequately from any toxicity and/or complications from the surgery before the first dose of study intervention
* Has a current stoma. Inclusion will be possible after continuity restoration (during the 5 weeks following continuity restoration)
* Has active anal fistula
* Is scheduled, according to SoC, to receive a biotherapy at the exception of anti-TNF agent in the 6 months after surgery
* Has had more than 2 past small bowel resections or cumulated intestinal resection superior to 50 cm
* Has a contraindication to endoscopy or anaesthesia.
* Is receiving antibiotics at time of randomization or is likely to require antibiotic treatment within 6 weeks of the first dose of EXL01 or placebo.
* Has a history of hypersensitivity to EXL01 and/or any excipients, which are listed in the Investigator Brochure (IB), and/or to soybean or soy-containing products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-09-13 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the distribution of endoscopic modified Rutgeerts scores, as centrally assessed, at 6 months post-surgery in patients with CD treated with EXL01 to patients treated with placebo. | From enrollment to the end of treatment at 24 weeks
  Evaluation of the distribution of modified Rutgeerts score grouped in 4 categories (i0: No lesions in the neoterminal ileum, i1: ≤ 5 ulcerations in the neoterminal ileum - i2a: Isolated anastomotic ulceration, i2b: >5 ulcerations in the neoterminal ileum, i3: Diffuse ileitis - i4: Diffuse ileitis with deep ulcerations and/or stenosis) at Week 24/EOT, evaluated by endoscopy with video capture, and assessed by BICR.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Allez, Principal Investigator — Remind
Locations (12):
- France (12):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU Lille, Lille
  - Hospices civils Lyon Sud, Lyon
  - CHU Marseille Nord, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice Archet 2, Nice
  - CHU Saint Louis, Paris
  - Hôpital Saint Antoine, Paris

IPD SHARING:
Plan to Share IPD: No